CLINICAL TRIAL: NCT07401459
Title: Multicenter Randomized Controlled Trial of a Multimodal AI Agent for Ophthalmology Clinical Decision Support
Brief Title: A Multimodal AI Agent for Ophthalmic Clinical Decision Support
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: PolyU-IRB-2025-001
Record Dates: First submitted 2025-11-17; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2025-09

CONDITIONS: Ophthalmology; Large Language Models; AI Agent; Eye Disease; Retinal Disease
Keywords: medical AI agent; large language model; ophthalmology; tool integration; clinical decision support; real world study
MeSH Terms: conditions — Eye Diseases; Retinal Diseases

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AI-assisted care arm (Experimental): Clinicians perform report generation, diagnosis, and treatment planning with support from the EyeAgent system.
  Interventions: Device: EyeAgent AI system
- Standard care arm (No Intervention): Clinicians provide routine ophthalmic care without support from the EyeAgent system.

INTERVENTIONS:
Device: EyeAgent AI system — EyeAgent is a multimodal AI agent assistant for ophthalmology that integrates imaging, electronic health records, and curated clinical knowledge. In this arm, EyeAgent supports clinicians in clinical consultation, including report generation, diagnostic interpretation, and treatment planning.
  Arms: AI-assisted care arm

SUMMARY:
This study is a multicenter randomized controlled trial evaluating the effectiveness and safety of EyeAgent, a multimodal artificial intelligence (AI) agent designed to assist ophthalmologists in clinical decision-making. Participants will be recruited from ophthalmology clinics and hospitals in Hong Kong and mainland China. The AI agent acts as a digital co-pilot, analyzing patient images and clinical history to provide diagnostic and management recommendations. The trial aims to determine whether the use of the AI agent improves diagnostic accuracy, treatment decision-making performance, report generation, workflow efficiency, and user satisfaction compared to standard clinical practice.

DETAILED DESCRIPTION:
This multicenter, randomized controlled trial aims to evaluate the integration of EyeAgent, a multimodal artificial intelligence (AI) agent, in real-world clinical settings. The AI system is designed to support clinicians by analyzing patient data, including ocular images and electronic health records, to aid in image interpretation, diagnosis, and treatment planning.

A total of 300 participants will be randomly assigned to either an AI-assisted care arm or a standard care arm. In the AI-assisted arm, clinicians review the comprehensive report generated by AI agent as a supportive tool before finalizing their independent decisions. The study comprehensively measures diagnostic accuracy, the rate of inappropriate treatment decisions, report generation, workflow efficiency, and user questionnaire.

By comparing these two groups, the trial aims to provide robust evidence on the effectiveness and practical utility of AI-driven clinical decision support in ophthalmology, with the goal of enhancing both the quality and efficiency of patient care.

ELIGIBILITY:
Inclusion Criteria:

1. Outpatient participants aged 6 to 75 years.
2. Participants who undergo ophthalmic examinations for medical purposes during the study period.
3. Participants who can produce clear ophthalmic images in both eyes.
4. Agree to participate in this study with written informed consent:

   1. Participants aged 18 years or older provide their own consent.
   2. Participants aged 6-17 years require consent from a parent or legal guardian.

Exclusion Criteria:

1. Participants who are reluctant to participate in this study.
2. Participants presenting with acute or emergency ocular conditions requiring immediate intervention.
3. Participants with poor quality of ophthalmic images, including blurriness, artifacts, underexposure, or overexposure.
4. Other unsuitable reasons determined by the evaluators.

Ages: 6 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy rate | Immediately after the intervention.
  Proportion of diagnoses consistent with a reference expert panel.
Rate of inappropriate treatment decisions | Immediately after the intervention.
  The frequency of treatment recommendations (e.g., injection, laser therapy, or observation) that deviate from clinical guidelines as determined by the senior expert panel gold standard. Expert adjudication is conducted post-hoc after the enrollment phase concludes.

SECONDARY OUTCOMES:
Report quality | Within 1 month after enrollment.
  Completeness and clarity of clinical reports, assessed via a standardized scoring rubric.
Clinician confidence | Immediately after the intervention.
  Clinician's self-rated confidence in diagnosis and treatment plans post-consultation.
Workflow efficiency | During the index diagnostic session.
  Time elapsed from image acquisition to final diagnosis and report completion.
Satisfaction and usability score | At the end of each clinician's participation period, approximately 2 months.
  Evaluation of the AI agent's user-friendliness, helpfulness, and logical transparency, measured via a structured 5-point Likert scale questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Mingguang He, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, China

IPD SHARING:
Plan to Share IPD: Undecided